CLINICAL TRIAL: NCT00072800
Title: Classification of Cerebral Palsy Subtypes
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040034; 04-N-0034
Record Dates: First submitted 2003-11-10; First posted 2003-11-11 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-08

CONDITIONS: Cerebral Palsy
Keywords: Reliability; Muscle Tone Abnormality; Spasticity; Dystonia; Rigidity; Cerebral Palsy; CP; Children
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity; Dystonia; Muscle Rigidity

SUMMARY:
This study, conducted at the National Institutes of Health and the Children's National Medical Center, will evaluate how well different physicians agree in how they classify cerebral palsy subtypes based on patient examination. Cerebral palsy is divided into several subtypes, according to the primary underlying muscle abnormality and its distribution and severity. Classification of these subtypes is important for conducting rehabilitation research studies on patients with the same type of abnormality. However, doctors do not always classify cerebral palsy types in the same way. This study will examine methods for improving agreement among doctors in their classification of cerebral palsy subtypes.

Children between 6 and 18 years of age with cerebral palsy who can voluntarily move their arms and legs may be eligible for this study. Participants will be examined by at least three doctors or therapists. The examinations take 30-60 minutes. For the examination, a doctor or therapist will do the following:

* Observe the patient at rest
* Gently move the patient's arms and legs and then have the patient move his or her arms and legs
* Check the patient's reflexes
* Observe the patient walking, if the patient is able to walk

Patients will be asked to remain in the clinic for up to 3 hours while researchers discuss the examination and may be asked to repeat part of the study examination.

DETAILED DESCRIPTION:
The movement and posture abnormalities that are characteristic of cerebral palsy are associated with underlying abnormalities of muscle tone, including dystonia, spasticity, and rigidity. The subtypes of cerebral palsy are defined according to the predominant muscle tone abnormality, its distribution and severity. There is widespread agreement that CP subtypes should be divided into the following groups. Spastic subtypes (hemiplegia: unilateral asymmetric spasticity; diplegia: bilateral symmetric spasticity, lower limbs more affected than upper limbs; quadriplegia: bilateral symmetric spasticity, upper and lower limbs affected equally), dystonic or athetotic type; and other miscellaneous types: hypotonic, mixed types, etc. These descriptive definitions are not useful when forming homogeneous cohorts of CP subtypes in rehabilitation research studies. Even when a preceding training session establishes precise criteria for each subtype based on these definitions and uses a "four limb" approach (defining the dominant muscle tone abnormality and its severity in each limb) the interobserver agreement in the classification of CP subtypes remains poor. This may be because there are no widely accepted definitions for the most common muscle tone abnormalities in cerebral palsy (spasticity, rigidity, dystonia) and examination methods vary widely. Recently, an interdisciplinary group of clinicians published a consensus document in which they set forth clear definitions for these disorders of muscle tone and recommendations on how to examine for them. Since the CP subtypes are defined according to the dominant muscle tone abnormality, we hypothesize that it may be possible to achieve acceptable interobserver agreement in the classification of the CP subtypes if these definitions and standard examination techniques are incorporated into the preceding training session with the other accepted elements. To test this hypothesis we will train clinicians from three different areas of expertise: child neurology, physiatry, physical therapy to classify subtypes of CP using accepted methods (establishing precise criteria for the subtypes and using a four limb approach) and will also train them to identify muscle tone abnormalities using the definitions and standard examination techniques in the consensus document. Following this training, we will ask the same clinicians to classify subtypes of cerebral palsy in a group of CP children. We will then measure interobserver agreement for the classification of CP using the kappa statistic. Achieving acceptable interobserver agreement in the classification of CP subtypes may facilitate the formation of homogeneous cohorts in research studies.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Children 6 to 18 years of age
2. Children must be previously diagnosed with cerebral palsy
3. Children born at any gestational age will be eligible.
4. Lesions must be pre-, peri- or post-natal and acquired before 2 years of age
5. Lesions must be non-progressive
6. Patients must be able to voluntarily move their upper and lower limbs

EXCLUSION CRITERIA:

1. Any subject who is pregnant
2. Children with an underlying known genetic or chromosomal disorder
3. Children with clearly identified familial or non-familial syndromes (without known chromosomal or genetic defect)
4. Cerebral lesions acquired after 2 years of age
5. Patients with progressive or neurodegenerative disorders
6. Patients with spinal disorders in the absence of cerebral lesions
7. Patients with sickle cell disease
8. Patients with cerebral lesions caused by emboli associated with congenital cardiac lesions
9. Patients with severe cognitive deficits who cannot follow simple verbal commands
10. Patients incapable of voluntary movement of either upper or lower limbs due to contractures.
11. Patients with prior rhizotomy
12. Patients with prior orthopedic (bone or soft tissue) surgery or serial casting
13. Patients with severe postural abnormalities who cannot maintain supported sitting.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115
Dates: Start 2003-11; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Sanger TD, Delgado MR, Gaebler-Spira D, Hallett M, Mink JW; Task Force on Childhood Motor Disorders. Classification and definition of disorders causing hypertonia in childhood. Pediatrics. 2003 Jan;111(1):e89-97. doi: 10.1542/peds.111.1.e89. PMID 12509602
- [Background] Colver AF, Sethumadhavan T. The term diplegia should be abandoned. Arch Dis Child. 2003 Apr;88(4):286-90. doi: 10.1136/adc.88.4.286. No abstract available. PMID 12651747
- [Background] Brashear A, Zafonte R, Corcoran M, Galvez-Jimenez N, Gracies JM, Gordon MF, McAfee A, Ruffing K, Thompson B, Williams M, Lee CH, Turkel C. Inter- and intrarater reliability of the Ashworth Scale and the Disability Assessment Scale in patients with upper-limb poststroke spasticity. Arch Phys Med Rehabil. 2002 Oct;83(10):1349-54. doi: 10.1053/apmr.2002.35474. PMID 12370866